CLINICAL TRIAL: NCT04257227
Title: Transcranial Magnetic Stimulation for Psychological Distress in Patients With Advanced Illness: A Phase 2a/2b Dose-finding and Feasibility Clinical Trial
Brief Title: Transcranial Magnetic Stimulation for Psychological Distress in Patients With Advanced Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Lotte & John Hecht Memorial Foundation (Other); Bruyère Health Research Institute. (Other); Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-19-035
Record Dates: First submitted 2019-12-11; First posted 2020-02-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Depressive Symptoms; Depression, Anxiety; Psychological Distress; Terminal Illness
Keywords: palliative care; end of life; repetitive transcranial magnetic stimulation; dose-finding; feasibility
MeSH Terms: conditions — Depression; Anxiety Disorders; Death | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Open-label dose-finding study, to be followed by either a sham-crossover or sham-control randomized clinical trial based on results of the dose-finding study. Study design described here is for the dose-finding study, and information will be updated once the randomized clinical trial is started.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rTMS Intervention Group (Experimental)
  Interventions: Device: repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation (rTMS) — The rTMS intervention will be performed in a dedicated rTMS patient room on the PC unit, where the patient can remain in their bed seated upwards at a 45 degree angle, or seated in a chair.
  The stimulation intensity for treatment will be determined by measuring the resting and active motor threshold (rMT and aMT) using single pulse TMS over the motor cortex using standard techniques as in previous trials. Investigators will use left-sided intermittent theta burst stimulation (iTBS). The trained team member will locate the left DLPFC using the BeamF3 technique. For the open-label dose-finding study, this region will be stimulated intermittently at 3 TMS pulses every 200 milliseconds for 2 seconds (i.e. 30 stimulations). This procedure is repeated every 10 seconds for a total duration of 3 minutes during which 600 total pulses are delivered. Participants will receive up to 8 3-minute sessions daily at 45 minute intervals for 5 days (consecutively or in a seven-day window if need be).
  Other Names: intermittent theta burst stimulation (iTBS)

SUMMARY:
Psychological and existential distress are a common cause of suffering among patients nearing the end of life, and a major reason for requesting medical aid in dying. Existing treatments for psychological and existential suffering have low efficacy and are challenging to use in a palliative context. There is a need to develop scalable, brief, and rapidly effective therapeutic approaches that can reduce psychological and existential distress in patients nearing the end of life.

Repetitive Transcranial Magnetic Stimulation is an effective treatment for refractory depression, and new protocols and increasing availability of rTMS may make this therapy feasible and acceptable for patients who suffer from psychological or existential distress near the end of life.

Among patients with advanced illness followed by a PC provider, the study objectives are to:

1. Identify the lowest and range of therapeutic rTMS dose to relieve psychological distress, including an analysis of clinical predictors of response.
2. Test the feasibility and preliminary efficacy of rTMS for the treatment of psychological distress including: 1) ease of recruitment; 2) completion of follow-up; 3) effect size and variance estimates of treatment for primary and secondary outcomes; and 4) patient satisfaction with treatment.

This study is a phase 2a dose-finding open-label clinical trial, followed by a phase 2b prospective, sham-control or sham-crossover study, depending on the therapeutic dose identified in phase 2a.

The investigators will enroll eligible patients from an inpatient palliative care unit and administer rTMS according to established best practice international guidelines. Two screening tests will be conducted (one completed by patient and another by the treating physician) to ensure the patient has no contraindications to rTMS. In the open-label dose-finding study, investigators will determine the appropriate dose of treatment that leads to positive patient outcomes, assess characteristics associated with positive and rapid response to rTMS, and examine if this treatment is feasible and acceptable to patients by measuring rates of enrollment and completion of the treatment sessions. Based on results from this first phase, a phase 2b feasibility and preliminary efficacy randomized clinical trial will be conducted to measure the effect of rTMS by comparing patient symptoms before and after the rTMS intervention.

DETAILED DESCRIPTION:
Patients with advanced illness often report feeling of depression and anxiety, struggling with loss of autonomy and relationships, a sense of hopelessness, and lack of meaning and purpose in life. These feelings have been described as "existential distress", and are associated with poor outcomes including decreased medication adherence, decreased quality of life, increased desire for hastened death, and increased rates of suicide. Existential distress, estimated to occur in up to 19% of patients with cancer nearing the end-of-life, has been identified as the primary reason why individuals pursue medical assistance in dying (MAiD), highlighting the impact existential and psychological suffering has on patients at the end-of-life.

There are few options for treating psychological or existential suffering in a palliative care (PC) population. Pharmacological approaches may reduce symptoms of depression and anxiety, but evidence to support the efficacy of antidepressants and anxiolytics is underwhelming. Antidepressant and anxiolytic medications may also take some time to show efficacy, and can cause serious side effects such as falls and confusion. The delayed effectiveness and potential for side effects can be substantial deterrents for many patients. Psychotherapeutic interventions can be used to reduce psychological suffering in patients with advanced illness, but results from randomized controlled trials have shown limited efficacy. Psychotherapy can be time consuming and slow to work, which is not ideal for patients with limited life expectancy. Given the burden of existential distress among patients followed by PC providers, there is a need to develop scalable, brief, and rapidly effective therapeutic approaches that can reduce existential distress in patients nearing the end-of-life.

Repetitive Transcranial Magnetic Stimulation (rTMS) is a Health-Canada- and FDA-approved safe and non-invasive brain stimulation intervention used to treat major depression, post-traumatic stress disorder, and other mood and anxiety disorders where medication has been ineffective. The technique uses trains of powerful, focused magnetic pulses, applied via a handheld inductor placed against the scalp, to induce changes in the activity of frontal lobe circuits responsible for regulating cognition and emotion. The most common stimulation protocols target the dorsolateral prefrontal cortex (DLPFC), using high-frequency (10-20 Hz) to the left DLPFC or low-frequency (1 Hz) to the right DLPFC, or both. With therapeutic rTMS, multiple sessions of treatment are delivered daily over 20-30 visits, to achieve durable symptomatic improvements. Clinical studies have shown rTMS can achieve a response (>50% symptom reduction) in half of patients and sustained remission rates in approximately 1/3 of patients whose depression has been refractory to 2 or more medications.

rTMS is generally well-tolerated with very few complications; about 95% of patients are able to complete a full course of treatment. However, there are obvious barriers to using traditional rTMS in the terminal population. First, the need to come to an rTMS clinic for a 60-minute session daily for 4-6 weeks is too great a time commitment for most patients nearing the end-of-life. Second, rTMS was only recently approved for public funding in many Canadian provinces, limiting the availability of rTMS to research settings and private clinics until now. Third, rTMS devices have been historically costly and difficult to transport, making it unfeasible for inpatient PC facilities to purchase an rTMS device or share one with a psychiatric clinic nearby. All of these factors have changed in the past couple years. New protocols of patterned rTMS have shortened treatment sessions yet preserve efficacy. Other "accelerated rTMS" protocols have given up to 10 sessions per day and shown symptom remission in just 2-5 days. The cost of these devices has also decreased dramatically in recent years (~$25,000 CAN), while the portability and availability have also improved, to the point that it is now feasible to use them in palliative settings.

The current body of literature presented above has studied the effectiveness of rTMS in patients with treatment-refractory depression and other mental illness. Essentially, the current treatment protocols have been designed to be effective in populations who are the most difficult to treat clinically. As such, there is no evidence as to whether or not patients with clinically less severe psychological distress (depression and anxiety), would require the same intensity and duration of treatment to achieve a clinically relevant therapeutic effect.

Objectives

Among patients with advanced illness followed by a PC provider:

1. Identify the lowest and range of therapeutic rTMS dose to relieve psychological distress, including an analysis of clinical predictors of response.
2. Test the feasibility and preliminary efficacy of accelerated rTMS for the treatment of psychological distress including: 1) ease of recruitment; 2) completion of follow-up; 3) effect size and variance estimates of treatment for primary and secondary outcomes; and 4) patient satisfaction with treatment.

Trial Design

The study is a phase 2a dose-finding open-label clinical trial, followed by a phase 2b prospective, sham-control or sham-crossover study, depending on the therapeutic dose identified in phase 2a.

Intervention and Control

The rTMS intervention will be performed in a dedicated rTMS patient room on an inpatient PC unit, where the patient can remain in their bed seated upwards at a 45 degree angle, or seated comfortably in a chair.

The stimulation intensity for the treatment will be determined by measuring the resting and active motor threshold (rMT and aMT) using single pulse TMS over the motor cortex using standard techniques as in previous trials. Investigators will use left-sided intermittent theta burst stimulation (iTBS) because it appears to achieve greater reductions in depressive symptoms and suicidal thoughts. The trained team member will locate the left DLPFC using the BeamF3 technique, which does not require neuroimaging and achieves comparably accurate positioning. For the phase 2a open-label dose-finding study, this region will be stimulated intermittently at 3 TMS pulses every 200 milliseconds for 2 seconds (i.e. 30 stimulations). This procedure is repeated every 10 seconds for 3 minutes during which 600 total pulses are delivered. Participants will receive up to 8 3-minutes sessions daily at 45 minute intervals for 5 days (consecutively or in a seven-day window if need be).

The results of this dose-finding study will inform the appropriate therapeutic dose to be provided to treatment-group participants in the phase 2b feasibility and preliminary efficacy trial. For example, if the dose-finding study demonstrates patients have a clinical response after just 3 days of treatment or 24 total doses, this will be the new treatment protocol for the phase 2b feasibility study.

For the sham intervention in the phase 2b feasibility and preliminary efficacy trial, the active coil will be replaced by a "sham" coil, which produces similar sound and scalp sensations as the active coils, but delivers no effective cortical stimulation.

Should the results of the dose-finding study demonstrate a low dose and minimal time is required to achieve therapeutic effect (e.g. 15 sessions over 3 days), the investigators will proceed with a sham-crossover study in which each patient will receive either the treatment or sham intervention first, followed by a 4-day washout period, after which they will receive either the treatment or sham intervention (whichever they did not receive the first round). Each patient thus serves as their own control. Alternatively, should the results demonstrate a high dose and time commitment (e.g. 40 sessions over 5 days) is required to achieve therapeutic effect, investigators will proceed with a sham-control design in which each patient will be randomized to receive either rTMS only or the sham control only. This decision is based on the rationale that it would be too cumbersome to ask patients to dedicate a minimum of 2 full weeks (5 days of treatment or sham, followed by a 4 day washout period, followed by another 5 days of treatment or sham) to this study, given these individuals are experiencing advanced illness.

Sample Size

To facilitate dose-finding in the phase 2a open-label trial, investigators will enroll patients until a clear threshold for therapeutic effect is identified, up to a maximum of 15 patients.

For the phase 2b feasibility and efficacy trial, investigators will aim to recruit 25 patients for the sham-crossover design, or 40 patients (n=20 treatment and n=20 control) for the sham-control design.

Recruitment

Each patient admitted to the PC unit will automatically be screened for eligibility by a research staff member and the treating PCU physician. Research staff will look at each newly admitted patient's Edmonton Symptom Assessment System (ESAS) score in the medical chart. A score of 7 or greater on the Depression, Anxiety or Well-being subscale of the ESAS will trigger research staff to approach the patient's physician to ensure the patient has an expected >1 month to live and is capable (physically and cognitively) of participating in the study. Both prospective participants and their physician will complete a screening questionnaire to ensure no contraindications to rTMS treatment.

Potential participants from the community will be identified by a member of their regional palliative care team (RPCT). A score of 7 or greater on the Depression, Anxiety or Well-being subscale of the ESAS and an expectation that the patient has an expected >1 month to live while being capable (physically and cognitively) of participating in the study will trigger an RPCT member to approach the patient to determine whether they are interested in the study. Both prospective participants and their health care provider will complete a screening questionnaire to ensure no contraindications to rTMS treatment.

For the phase 2b feasibility and preliminary efficacy trial, controls will be recruited in the same manner.

Allocation and Blinding

Investigators will use a random sequence generator for clinical trials. Information about allocation sequence will only be available to the trained research staff member who is administering the rTMS.

During the phase 2b feasibility and preliminary efficacy clinical trial, participants will be randomized to treatment versus sham (either order of treatment vs. sham is randomized in a sham-crossover, or the receipt of treatment or sham is randomized in a sham-control design). Participants will not be made aware of their randomization status and treatment allocation (i.e. participant blinding).

Study investigators will also be blinded to intervention allocation. The only individual who will have knowledge of the participant's intervention allocation is the trained rTMS operator who will be delivering the intervention.

Statistical Methods

Analysis of study results for the dose-finding study will be descriptive and correlational. Investigators will use descriptive statistics to examine the characteristics of participants who had a positive response to rTMS/ responded the quickest compared to the characteristics of participants who did not respond to rTMS treatment/had a slower response. We will also use descriptive measures (mean, median and respective confidence estimates) to evaluate the dose when 50% of participants, for example, experienced an improvement in symptoms.

Main analyses for the feasibility outcomes in both the dose-finding and phase 2b trial study will include calculation of outcomes using descriptive statistics with 95% confidence intervals. As the main aim is one of estimation rather than hypothesis testing, variance estimates and effect sizes with 95% confidence intervals will be calculated for primary and secondary efficacy measures in favour of significance testing.

Analysis for the phase 2b trial specifically will adopt an intention to treat approach. Assessment for a crossover effect should we use a sham-crossover design will employ a statistical analysis comparing the change in symptoms from before to after treatment in each patient over the sham period versus the active period. Assessment for a between-groups difference will be done should a sham-control design be employed.

ELIGIBILITY:
Inclusion Criteria:

* PC unit patients and PC patients in the community with advanced (terminal) illness
* >1 month life expectancy
* Experiencing psychological distress, as indicated by a score of 7 or greater on the Depression, Anxiety, or Well-being subscale of the Edmonton Symptom Assessment System (ESAS)
* Ability to understand and communicate in English

Exclusion Criteria:

* Current or previously diagnosed seizure disorder or first-degree relative with current or previously diagnosed seizure disorder
* Documented brain lesions
* Inability to remain still while sitting up (45 degrees) for the duration of therapy
* Known contraindications to rTMS, including: metallic skull plates, clips, or stimulators; pacemakers and other electronic implants; pregnancy; recurrent headaches with no known cause that do not respond to over-the-counter medications; current or previous skull fracture or traumatic brain injury; previous brain surgery; medications that lower seizure threshold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Change in Psychological Distress, Depression | Baseline (1 day prior to treatment start); after each day of rTMS treatment; 2 weeks, 4, and 8 weeks after intervention completion, if participant is alive
  17-Item Hamilton Rating Scale for Depression (HRSD); scores 0-52; higher score is more severe depression
Change in Psychological Distress, Depression and Anxiety | Baseline (1 day prior to treatment start); after each day of rTMS treatment; 2 weeks, 4, and 8 weeks after intervention completion, if participant is alive
  The Hospital Anxiety and Depression Scale (HADS); scores 0-21; higher score is more severe anxiety/depression
Recruitment Rate | Measured upon study enrollment termination (estimated at 8 months for dose-finding study)
  Total number of participants divided by the total number of eligible patients approached
Recruitment Rate | Measured upon study enrollment termination (estimated at 12 months for feasibility randomized clinical trial)
  Total number of participants divided by the total number of eligible patients approached
Completion of Intervention | Through intervention completion, up to 1 week
  The total number of rTMS sessions completed per day (maximum 8 sessions/day)
Completion of Intervention | Last day of rTMS treatment, at treatment day 5
  The total number of days of rTMS treatment received (maximum 5 days)
Completion of Follow-up | Upon study completion (up to 20 months)
  Proportion of enrolled participants who complete all assessments at 2 weeks, 4 weeks, and 8 weeks post-intervention

SECONDARY OUTCOMES:
Anxiety | Baseline (1 day prior to treatment start); end of last rTMS treatment day; 2 weeks, 4 weeks, 8 weeks, and 3 months after intervention completion, if participant is alive
  Hamilton Rating Scale for Anxiety; scores 0-30; higher score is more severe anxiety
Existential Distress | Baseline (1 day prior to treatment start); end of last rTMS treatment day; 2 weeks, 4 weeks, 8 weeks, and 3 months after intervention completion, if participant is alive
  24-Item Demoralization (DEM) Scale; scores 0-96; higher score is more severe demoralization
Death Anxiety | Baseline (1 day prior to treatment start); end of last rTMS treatment day; 2 weeks, 4 weeks, 8 weeks, and 3 months after intervention completion, if participant is alive
  Revised Death Anxiety Scale (RDAS) score; scores 15-75; higher score is more severe death anxiety
Participant Quality of Life: WHOQOL-Bref | Baseline (1 day prior to treatment start); end of last rTMS treatment day; 2 weeks, 4 weeks, 8 weeks, and 3 months after intervention completion, if participant is alive
  World Health Organization Quality of Life Scale-brief version (WHOQOL-Bref); transformed scores range 4-20; higher score is higher quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Elisabeth Bruyère Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauereiss N, Obermaier S, Ozunal SE, Baumeister H. Effects of existential interventions on spiritual, psychological, and physical well-being in adult patients with cancer: Systematic review and meta-analysis of randomized controlled trials. Psychooncology. 2018 Nov;27(11):2531-2545. doi: 10.1002/pon.4829. Epub 2018 Aug 2. PMID 29958339
- [Background] Arrieta O, Angulo LP, Nunez-Valencia C, Dorantes-Gallareta Y, Macedo EO, Martinez-Lopez D, Alvarado S, Corona-Cruz JF, Onate-Ocana LF. Association of depression and anxiety on quality of life, treatment adherence, and prognosis in patients with advanced non-small cell lung cancer. Ann Surg Oncol. 2013 Jun;20(6):1941-8. doi: 10.1245/s10434-012-2793-5. Epub 2012 Dec 22. PMID 23263699
- [Background] Colleoni M, Mandala M, Peruzzotti G, Robertson C, Bredart A, Goldhirsch A. Depression and degree of acceptance of adjuvant cytotoxic drugs. Lancet. 2000 Oct 14;356(9238):1326-7. doi: 10.1016/S0140-6736(00)02821-X. PMID 11073026
- [Background] Skarstein J, Aass N, Fossa SD, Skovlund E, Dahl AA. Anxiety and depression in cancer patients: relation between the Hospital Anxiety and Depression Scale and the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire. J Psychosom Res. 2000 Jul;49(1):27-34. doi: 10.1016/s0022-3999(00)00080-5. PMID 11053601
- [Background] Bovero A, Sedghi NA, Opezzo M, Botto R, Pinto M, Ieraci V, Torta R. Dignity-related existential distress in end-of-life cancer patients: Prevalence, underlying factors, and associated coping strategies. Psychooncology. 2018 Nov;27(11):2631-2637. doi: 10.1002/pon.4884. Epub 2018 Sep 24. PMID 30189464
- [Background] Li M, Watt S, Escaf M, Gardam M, Heesters A, O'Leary G, Rodin G. Medical Assistance in Dying - Implementing a Hospital-Based Program in Canada. N Engl J Med. 2017 May 25;376(21):2082-2088. doi: 10.1056/NEJMms1700606. No abstract available. PMID 28538128
- [Background] Hendry M, Pasterfield D, Lewis R, Carter B, Hodgson D, Wilkinson C. Why do we want the right to die? A systematic review of the international literature on the views of patients, carers and the public on assisted dying. Palliat Med. 2013 Jan;27(1):13-26. doi: 10.1177/0269216312463623. Epub 2012 Nov 5. PMID 23128904
- [Background] Salt S, Mulvaney CA, Preston NJ. Drug therapy for symptoms associated with anxiety in adult palliative care patients. Cochrane Database Syst Rev. 2017 May 18;5(5):CD004596. doi: 10.1002/14651858.CD004596.pub3. PMID 28521070
- [Background] Lo C, Hales S, Jung J, Chiu A, Panday T, Rydall A, Nissim R, Malfitano C, Petricone-Westwood D, Zimmermann C, Rodin G. Managing Cancer And Living Meaningfully (CALM): phase 2 trial of a brief individual psychotherapy for patients with advanced cancer. Palliat Med. 2014 Mar;28(3):234-42. doi: 10.1177/0269216313507757. Epub 2013 Oct 29. PMID 24170718
- [Background] Chochinov HM, Kristjanson LJ, Breitbart W, McClement S, Hack TF, Hassard T, Harlos M. Effect of dignity therapy on distress and end-of-life experience in terminally ill patients: a randomised controlled trial. Lancet Oncol. 2011 Aug;12(8):753-62. doi: 10.1016/S1470-2045(11)70153-X. Epub 2011 Jul 6. PMID 21741309
- [Background] Downar J, Blumberger DM, Daskalakis ZJ. Repetitive transcranial magnetic stimulation: an emerging treatment for medication-resistant depression. CMAJ. 2016 Nov 1;188(16):1175-1177. doi: 10.1503/cmaj.151316. Epub 2016 Aug 22. No abstract available. PMID 27551033
- [Background] Tik M, Hoffmann A, Sladky R, Tomova L, Hummer A, Navarro de Lara L, Bukowski H, Pripfl J, Biswal B, Lamm C, Windischberger C. Towards understanding rTMS mechanism of action: Stimulation of the DLPFC causes network-specific increase in functional connectivity. Neuroimage. 2017 Nov 15;162:289-296. doi: 10.1016/j.neuroimage.2017.09.022. Epub 2017 Sep 12. PMID 28912081
- [Background] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Background] Brunelin J, Jalenques I, Trojak B, Attal J, Szekely D, Gay A, Januel D, Haffen E, Schott-Pethelaz AM, Brault C; STEP Group; Poulet E. The efficacy and safety of low frequency repetitive transcranial magnetic stimulation for treatment-resistant depression: the results from a large multicenter French RCT. Brain Stimul. 2014 Nov-Dec;7(6):855-63. doi: 10.1016/j.brs.2014.07.040. Epub 2014 Aug 7. PMID 25192980
- [Background] McGirr A, Van den Eynde F, Tovar-Perdomo S, Fleck MP, Berlim MT. Effectiveness and acceptability of accelerated repetitive transcranial magnetic stimulation (rTMS) for treatment-resistant major depressive disorder: an open label trial. J Affect Disord. 2015 Mar 1;173:216-20. doi: 10.1016/j.jad.2014.10.068. Epub 2014 Nov 11. PMID 25462419
- [Background] Fitzgerald PB, Hoy KE, Elliot D, Susan McQueen RN, Wambeek LE, Daskalakis ZJ. Accelerated repetitive transcranial magnetic stimulation in the treatment of depression. Neuropsychopharmacology. 2018 Jun;43(7):1565-1572. doi: 10.1038/s41386-018-0009-9. Epub 2018 Feb 5. PMID 29467437
- [Background] Baeken C, Marinazzo D, Wu GR, Van Schuerbeek P, De Mey J, Marchetti I, Vanderhasselt MA, Remue J, Luypaert R, De Raedt R. Accelerated HF-rTMS in treatment-resistant unipolar depression: Insights from subgenual anterior cingulate functional connectivity. World J Biol Psychiatry. 2014 May;15(4):286-97. doi: 10.3109/15622975.2013.872295. Epub 2014 Jan 21. PMID 24447053
- [Background] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360
- [Background] Fitzgerald PB, Hoy K, Gunewardene R, Slack C, Ibrahim S, Bailey M, Daskalakis ZJ. A randomized trial of unilateral and bilateral prefrontal cortex transcranial magnetic stimulation in treatment-resistant major depression. Psychol Med. 2011 Jun;41(6):1187-96. doi: 10.1017/S0033291710001923. Epub 2010 Oct 7. PMID 20925972
- [Background] Cooper YA, Pianka ST, Alotaibi NM, Babayan D, Salavati B, Weil AG, Ibrahim GM, Wang AC, Fallah A. Repetitive transcranial magnetic stimulation for the treatment of drug-resistant epilepsy: A systematic review and individual participant data meta-analysis of real-world evidence. Epilepsia Open. 2017 Dec 27;3(1):55-65. doi: 10.1002/epi4.12092. eCollection 2018 Mar. PMID 29588988
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Kissane DW, Wein S, Love A, Lee XQ, Kee PL, Clarke DM. The Demoralization Scale: a report of its development and preliminary validation. J Palliat Care. 2004 Winter;20(4):269-76. PMID 15690829
- [Background] Templer DI. The construction and validation of a Death Anxiety Scale. J Gen Psychol. 1970 Apr;82(2d Half):165-77. doi: 10.1080/00221309.1970.9920634. No abstract available. PMID 4394812
- [Background] 46. World Health Organization. WHOQOL-BREf: Introduction, administration, scoring, and generic version of the assessment. Dec 1996. Retrieved from: https://www.who.int/mental_health/media/en/76.pdf
- [Background] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Derived] Downar J, Lapenskie J, Anderson K, Edwards J, Watt C, Dionne M, Rice J, Kabir M, Lawlor P, Downar J. Accelerated transcranial magnetic stimulation for psychological distress in advanced cancer: A phase 2a feasibility and preliminary efficacy clinical trial. Palliat Med. 2024 Apr;38(4):485-491. doi: 10.1177/02692163241234799. Epub 2024 Mar 14. PMID 38482823